CLINICAL TRIAL: NCT03845166
Title: A Dose-Escalation and Expansion Study of the Safety and Pharmacokinetics of XL092 as Single-Agent and Combination Therapy in Subjects With Inoperable Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of XL092 as Single-Agent and Combination Therapy in Subjects With Solid Tumors
Acronym: STELLAR-001
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XL092-001; 2020-003569-21 (EudraCT Number)
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Neoplasm Malignant; Renal Cell Carcinoma; Hormone Receptor Positive Breast Carcinoma; Metastatic Castration-resistant Prostate Cancer; Colorectal Cancer
MeSH Terms: conditions — Neoplasms; Carcinoma, Renal Cell; Colorectal Neoplasms | interventions — atezolizumab; avelumab

STUDY DESIGN:
Intervention Model Description: single-agent and combination therapy dose-escalation followed by cohort-expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- XL092 Single-Agent Dose-Escalation Cohorts (Experimental): Subjects will accrue in cohorts of 3-6 subjects in a standard "3 plus 3" design.
  Interventions: Drug: XL092
- XL092 Single-Agent Expansion Cohorts (Experimental): The MTD or recommended dose from the dose-escalation stage may be further explored in clear cell renal cell carcinoma (ccRCC), non-clear cell renal cell carcinoma (nccRCC), hormone receptor-positive breast cancer (HR+ BC), and metastatic castration-resistant prostate cancer (mCRPC).
  Interventions: Drug: XL092
- XL092 + Atezolizumab Dose-Escalation Cohorts (Experimental): Subjects will accrue in cohorts of 2-6 subjects in a "rolling 6" design.
  Interventions: Drug: XL092; Drug: Atezolizumab
- XL092 + Atezolizumab Expansion Cohorts (Experimental): The MTD or recommended dose from the dose-escalation stage may be further explored in non-clear cell renal cell carcinoma (nccRCC), hormone receptor-positive breast cancer (HR+ BC), metastatic castration-resistant prostate cancer (mCRPC), and colorectal cancer (CRC).
  Interventions: Drug: XL092; Drug: Atezolizumab
- XL092 + Avelumab Dose-Escalation Cohorts (Experimental): Subjects will accrue in cohorts of 2-6 subjects in a "rolling 6" design.
  Interventions: Drug: XL092; Drug: Avelumab

INTERVENTIONS:
Drug: XL092 — oral doses of XL092
Drug: Atezolizumab — Supplied as 1200 mg/20 mL vials; administered as a 1200 mg IV infusion once every 3 weeks (q3w)
  Other Names: Tecentriq®
  Arms: XL092 + Atezolizumab Dose-Escalation Cohorts; XL092 + Atezolizumab Expansion Cohorts
Drug: Avelumab — Supplied as 200 mg/10 mL vials; administered as an 800 mg IV infusion once every 2 weeks (q2w)
  Other Names: Bavencio®
  Arms: XL092 + Avelumab Dose-Escalation Cohorts

SUMMARY:
This is a Phase 1, open-label, dose-escalation and expansion study, evaluating the safety, tolerability, pharmacokinetics (PK), preliminary antitumor activity, and effect on biomarkers of XL092 administered alone, in combination with atezolizumab, and in combination with avelumab to subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed solid tumor that is inoperable locally advanced, metastatic, or recurrent.
* Dose-escalation (single-agent and combination therapy): Subjects with a solid tumor that is unresectable or metastatic and for which life-prolonging therapies do not exist or available therapies are intolerable or no longer effective.
* Expansion Cohort A (ccRCC): Subjects with previously treated advanced RCC with clear cell histology (including those with a sarcomatoid component) who have radiographically progressed following treatment with at least one prior systemic anticancer regimen for inoperable locally advanced or metastatic disease.
* Expansion Cohorts B and E (nccRCC): Subjects with previously treated advanced RCC with non-clear cell histology who have radiographically progressed following treatment with at least one prior systemic anticancer regimen for inoperable locally advanced or metastatic disease.
* Expansion Cohorts C and F (HR+ BC): Subjects with breast cancer that is hormone receptor positive (ER+ and/or PR+) and negative for human epidermal growth factor receptor 2 (HER-2) and who have radiographically progressed during or following treatment with at least one prior systemic anticancer regimen for inoperable locally advanced or metastatic disease.
* Expansion Cohorts D and G (mCRPC): Subjects with metastatic CRPC (adenocarcinoma of the prostate). Neuroendocrine differentiation and other features permitted if adenocarcinoma is the primary histology.
* Expansion Cohort H (CRC): Subjects with histologically confirmed unresectable, locally advanced, or metastatic adenocarcinoma of the colon or rectum, KRAS/NRAS wild-type (confirmed via local testing report) and determined NOT to have microsatellite instability high (MSI-high) or mismatch repair deficient (dMMR) by local testing, who received the following standard of care chemotherapy regimens as prior therapy for metastatic CRC:

  * Fluoropyrimidine, irinotecan and oxaliplatin, with or without an anti-VEGF monoclonal antibody (bevacizumab)
  * Anti-EGFR monoclonal antibody (cetuximab or panitumumab)
  * BRAF inhibitor (in combination with cetuximab +/- binimetinib) for subjects with BRAF V600E mutations
* Expansion Cohorts: Subjects must have measurable disease per RECIST 1.1.
* Tumor tissue material:

  * Subjects in the non-biomarker cohort provide archival, if available, or fresh tumor tissue if it can be safely obtained.
* Recovery to baseline or ≤ Grade 1 severity (CTCAE v5) from adverse events (AEs), including immune-related adverse events (irAEs), related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
* Adequate organ and marrow function.
* Sexually active fertile subjects and their partners must agree to use highly effective methods of contraception.
* Female subjects of childbearing potential must not be pregnant at screening.

Exclusion Criteria:

* Prior treatment with XL092 (all cohorts), prior treatment with PD-L1/PD-1 targeting immune checkpoint inhibitor (Cohorts E, F, G, and H only), or prior treatment with regorafenib and/or TAS-102 (Cohort H only).
* Receipt of any type of small molecule kinase inhibitor within 2 weeks before first dose of study treatment.
* Receipt of any type of anticancer antibody, systemic chemotherapy, or hormonal anticancer therapy within 4 weeks before first dose of study treatment.
* Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment.
* Uncontrolled, significant intercurrent or recent illness.
* Concomitant use of certain medications.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 450 ms for males and > 470 ms for females. Single ECGs are no longer permitted.
* Pregnant or lactating females.
* Diagnosis of another malignancy within 2 years before first dose of study treatment, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy.

Additional Exclusion Criteria for XL092 + Atezolizumab Combination Therapy Cohorts ONLY:

* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 2 weeks prior to first dose of study treatment.
* Administration of a live, attenuated vaccine within 30 days before first dose of study treatment.

Additional Exclusion Criteria for XL092 + Avelumab Combination Therapy Cohorts ONLY:

* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent.
* Administration of a live, attenuated vaccine within 30 days before first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Dose-Escalation Stage: MTD/recommended dose for XL092 | Up to 24 months
  To determine the maximum tolerated dose (MTD) and/or recommended dose (RD) for further evaluation of XL092 when administered alone and in combination with immune checkpoint inhibitors (ICIs) to subjects with advanced solid tumors
Cohort-Expansion Stage: Objective Response Rate (ORR) | Up to 24 months
  To evaluate preliminary efficacy of XL092 when administered alone and in combination with ICIs by estimating ORR as assessed by the Investigator per RECIST 1.1
Cohort-Expansion Stage (except Cohort H): Progression-Free Survival (PFS) | Up to 24 months
  To evaluate preliminary efficacy of single-agent XL092 and XL092 in combination with ICIs for specific cohorts by estimating the percentage of subjects with PFS at 6 months (PFS rate) per RECIST 1.1 as assessed by the Investigator (except for the CRC expansion cohort H)
Cohort-Expansion Stage (Cohort H only): Overall Survival (OS) | Up to 24 months
  To evaluate preliminary efficacy of single-agent XL092 and XL092 in combination with atezolizumab for subjects with RAS wild-type CRC (Cohort H Treatment Arms H-A and H-B) by estimating overall survival (OS)

SECONDARY OUTCOMES:
Incidence and Severity of Nonserious Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 36 months
  To evaluate the safety of XL092 when administered alone and in combination with ICIs through the evaluation of incidence and severity of nonserious AEs and SAEs, including immune-related adverse events (irAEs), and adverse events of special interest (AESIs)
Dose-Escalation Stage: Time to Maximum Plasma Concentration (Tmax) | Up to 24 months
  To evaluate the Tmax of XL092 alone and in combination with ICI
Dose-Escalation Stage: Maximum Plasma Concentration (Cmax) | Up to 24 months
  To evaluate the Cmax of XL092 alone and in combination with ICI
Dose-Escalation Stage: Area Under the Plasma Concentration-Time Curve Over the Last 24-hour Dosing Interval (AUC 0-24) | Up to 24 months
  To evaluate the AUC 0-24 of XL092 alone and in combination with ICI
Dose-Escalation Stage: Terminal Half-Life | Up to 24 months
  To evaluate the terminal half-life of XL092 alone and in combination with ICI
Dose-Escalation Stage: Apparent Clearance (CL/F) | Up to 24 months
  To evaluate the CL/F of XL092 alone and in combination with ICI

CONTACTS AND LOCATIONS:
Locations (86):
- United States (40):
  - Exelixis Clinical Site #6, Duarte, California
  - Exelixis Clinical Site #49, La Jolla, California
  - Exelixis Clinical Site #7, Los Angeles, California
  - Exelixis Clinical Site #84, Los Angeles, California
  - Exelixis Clinical Site #66, San Francisco, California
  - Exelixis Clinical Site #71, Stanford, California
  - Exelixis Clinical Site #15, Lake Mary, Florida
  - Exelixis Clinical Site #24, Miami, Florida
  - Exelixis Clinical Site #11, Atlanta, Georgia
  - Exelixis Clinical Site #80, Atlanta, Georgia
  - Exelixis Clinical Site #41, Iowa City, Iowa
  - Exelixis Clinical Site #36, Westwood, Kansas
  - Exelixis Clinical Site #62, Scarborough, Maine
  - Exelixis Clinical Site #44, Baltimore, Maryland
  - Exelixis Clinical Site #4, Boston, Massachusetts
  - Exelixis Clinical Site #45, Ann Arbor, Michigan
  - Exelixis Clinical Site #2, Grand Rapids, Michigan
  - Exelixis Clinical Site #25, Saint Paul, Minnesota
  - Exelixis Clinical Site #13, Omaha, Nebraska
  - Exelixis Clinical Site #9, East Brunswick, New Jersey
  - Exelixis Clinical Site #83, New Brunswick, New Jersey
  - Exelixis Clinical Site #86, New York, New York
  - Exelixis Clinical Site #35, New York, New York
  - Exelixis Clinical #78, New York, New York
  - Exelixis Clinical Site #85, The Bronx, New York
  - Exelixis Clinical #74, Cincinnati, Ohio
  - Exelixis Clinical Site #60, Cleveland, Ohio
  - Exelixis Clinical Site #59, Hershey, Pennsylvania
  - Exelixis Clinical Site #58, Philadelphia, Pennsylvania
  - Exelixis Clinical Site #12, Pittsburgh, Pennsylvania
  - Exelixis Clinical Site #61, Charleston, South Carolina
  - Exelixis Clinical Site #50, Myrtle Beach, South Carolina
  - Exelixis Clinical Site #33, Germantown, Tennessee
  - Exelixis Clinical Site #87, Nashville, Tennessee
  - Exelixis Clinical Site #3, Houston, Texas
  - Exelixis Clinical Site #1, San Antonio, Texas
  - Exelixis Clinical Site #5, Salt Lake City, Utah
  - Exelixis Clinical Site #8, Charlottesville, Virginia
  - Exelixis Clinical Site #43, Richmond, Virginia
  - Exelixis Clinical Site #26, Spokane, Washington
- Australia (5):
  - Exelixis Clinical Site #52, Darlinghurst, New South Wales
  - Exelixis Clinical Site #53, Liverpool, New South Wales
  - Exelixis Clinical #75, South Brisbane, Queensland
  - Exelixis Clinical Site #56, Kurralta Park, South Australia
  - Exelixis Clinical Site #63, Heidelberg, Victoria
- Belgium (3):
  - Exelixis Clinical Site #44, Edegem, Antwerpen
  - Exelixis Clinical Site #65, Ghent, Oost-Vlaanderen
  - Exelixis Clinical Site #51, Brussels
- Czechia (4):
  - Exelixis Clinical Site #21, Brno
  - Exelixis Clinical Site #42, Hradec Králové
  - Exelixis Clinical Site #10, Olomouc
  - Exelixis Clinical Site #27, Prague
- France (11):
  - Exelixis Clinical Site #46, Clermont, Ferrand
  - Exelixis Clinical Site #37, Saint-Herblain, Loire Atlantique
  - Exelixis Clinical #72, Bordeaux
  - Exelixis Clinical Site #32, Caen
  - Exelixis Clinical Site #48, Marseille
  - Exelixis Clinical Site #14, Paris
  - Exelixis Clinical Site #39, Pierre-Bénite
  - Exelixis Clinical Site #47, Poitiers
  - Exelixis Clinical Site #22, Suresnes
  - Exelixis Clinical Site #57, Toulouse
  - Exelixis Clinical #77, Villejuif
- Germany (3):
  - Exelixis Clinical Site #38, Nürtingen, Baden-Wurttemberg
  - Exelixis Clinical Site #31, Münster, North Rhine-Westphalia
  - Exelixis Clinical Site #64, Hamburg
- Italy (4):
  - Exelixis Clinical Site #67, Milan, MI
  - Exelixis Clinical Site #69, Pavia, PV
  - Exelixis Clinical Site #54, Milan
  - Exelixis Clinical #73, Napoli
- Netherlands (2):
  - Exelixis Clinical Site #79, Amsterdam, North Holland
  - Exelixis Clinical #76, Rotterdam, South Holland
- Spain (11):
  - Exelixis Clinical Site #23, Sabadell, Barcelona
  - Exelixis Clinical Site #20, Santiago de Compostela, La Coruna
  - Exelixis Clinical Site #18, Barcelona
  - Exelixis Clinical Site #19, Barcelona
  - Exelixis Clinical Site #29, Barcelona
  - Exelixis Clinical Site #30, Barcelona
  - Exelixis Clinical Site #81, Madrid
  - Exelixis Clinical Site #34, Madrid
  - Exelixis Clinical Site #55, Madrid
  - Exelixis Clinical Site #17, Madrid
  - Exelixis Clinical Site #16, Seville
- United Kingdom (3):
  - Exelixis Clinical #70, London, England
  - Exelixis Clinical Site #40, Sutton, England
  - Exelixis Clinical Site #68, Preston, Lancashire